CLINICAL TRIAL: NCT01676896
Title: Enhancing Children's and Parents' Asthma Management
Brief Title: Asthma in Central Texas Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: R01NR007770 (NIH); R01NR007770 (NIH)
Record Dates: First submitted 2012-08-24; First posted 2012-08-31 (Estimated); Results first posted 2015-04-02 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Asthma
Keywords: children; asthma; quality of life; self-management
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Asthma in-school class (Experimental): Provided in 16 15-minute sessions (4 hours total didactic time); scheduled 3 sessions/week. The content is provided by trained asthma educators. The Asthma Plan for Kids (AP-K) is a 7-step curriculum for children to use when responding to asthma symptoms. Skills practice with placebo metered dose inhaler (MDI) and peak expiratory flow (PEF) meters with PEF score interpretation. Topics include (a) identifying lung function, asthma warning signs, symptoms, and triggers; (b) learning skills to manage symptoms, including PEF meter score interpretation, communication with adults (e.g. teachers, coaches, family members), medication use and MDI technique; (c) evaluating asthma symptoms and the effectiveness of management; and (d) discussing how to stay active in a safe manner.
  Interventions: Behavioral: Asthma in-school class
- Asthma Day Camp (Experimental): The asthma day camp is provided in a single day session (5.5 hours total) by trained camp staff. The same skills (i.e., placebo metered dose inhaler (MDI) and peak expiratory flow (PEF) meters) and topics [a) identifying lung function, asthma warning signs, symptoms, and triggers; (b) learning skills to manage symptoms, including PEF meter score interpretation, communication with adults (e.g. teachers, coaches, family members), medication use and MDI technique; (c) evaluating asthma symptoms and the effectiveness of management; and (d) discussing how to stay active in a safe manner] are covered as those in the asthma in-school classes.
  Interventions: Behavioral: Asthma Day Camp
- Health Promotion in-school class (Sham Comparator): The mock comparison follows the in-school format of 16 15-minute sessions; scheduled 3 sessions/week. The content is provided by trained health educators and includes skills practice (i.e., handwashing and brushing teeth) and health promotion topics of nutrition, healthy snacks, preventing colds, and safe exercise.
  Interventions: Behavioral: Health Promotion in-school class

INTERVENTIONS:
Behavioral: Asthma in-school class
  Other Names: Asthma Plan for Kids
  Arms: Asthma in-school class
Behavioral: Asthma Day Camp
  Arms: Asthma Day Camp
Behavioral: Health Promotion in-school class
  Arms: Health Promotion in-school class

SUMMARY:
Asthma is the most common chronic childhood illness and disproportionately affects children who are ethnic minorities and poor. Few studies of childhood asthma have been conducted with children who live in rural areas or have included Mexican American children in their samples. This study builds on the original R01NR007770 with findings that demonstrated the intervention could improve children's asthma self-management, asthma knowledge, metered dose inhaler skill, asthma severity, and parents' asthma management and access to care. In this competing continuation, the investigators added a third arm to the current research design with schools randomized into either an in-school asthma intervention, an in-school attention-control intervention, or an alternate intervention-delivery format of a single 5.5-hour asthma day camp. The tri-ethnic sample will be composed of 320 Mexican-American, African-American, and White rural school-aged children (grades 2-5) who have asthma and their parents. In addition, the investigators propose adding a non-invasive measure of chronic airway inflammation (exhaled nitric oxide) to assess the impact of changes in asthma management on airway inflammation. Families will be followed for a full year with data collection at baseline and at 1-month, 4-months, and 7-months after the intervention to assess improvement in children's asthma morbidity, asthma severity, airway inflammation, family asthma management and quality of life. Hypotheses (H): Children in the Camp-Workshop group and the School-Home group will demonstrate equivalent improvements, but greater improvements than the Attention-Control group in:(H1.1) their asthma severity and airway inflammation from the Time 1 assessment when compared to Time 4 assessment; (H1.2) office visits, ED visits, and hospitalizations for asthma, and absenteeism for the study year (Time 4) when compared to the pre-study year (Time 1); and (H1.4) Parents in the intervention arms will demonstrate sustained improvements in asthma caregiver's quality of life (QOL0 from the pre-study year (Time 1) to the end of the study year (Time 4) measurement, when compared to the Attention-Control group.

DETAILED DESCRIPTION:
Families are recruited at the beginning of the school year (Time 1, October-November); parents consent and child assent obtained and baseline data collected in fall. The intervention is provided in December-January. Follow-up data are collected at February (Time 2), April (Time 3), and August (Time 4).

ELIGIBILITY:
Inclusion Criteria:

* parent reports the child has a diagnosis of asthma made by a medical provider;
* has had asthma symptoms in the previous 12 months;
* speaks either English or Spanish.

Exclusion Criteria:

* has a significant co-morbidity that would preclude participation in classes (e.g., severe cerebral palsy, oxygen dependent conditions)

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 292 (Actual)
Dates: Start 2008-12; Primary Completion 2013-09 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Texas at Austin, Austin, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Asthma In-school Class: Provided in 16 15-minute sessions (4 hours total didactic time); scheduled 3 sessions/week. The content is provided by trained asthma educators. The Asthma Plan for Kids (AP-K) is a 7-step curriculum for children to use when responding to asthma symptoms. Skills practice with placebo metered dose inhaler (MDI) and peak expiratory flow (PEF) meters with PEF score interpretation. Topics include (a) identifying lung function, asthma warning signs, symptoms, and triggers; (b) learning skills to manage symptoms, including PEF meter score interpretation, communication with adults (e.g. teachers, coaches, family members), medication use and MDI technique; (c) evaluating asthma symptoms and the effectiveness of management; and (d) discussing how to stay active in a safe manner.
  Asthma in-school class
- Asthma Day Camp: The asthma day camp is provided in a single day session (5.5 hours total) by trained camp staff. The same skills (i.e., placebo metered dose inhaler (MDI) and peak expiratory flow (PEF) meters) and topics [a) identifying lung function, asthma warning signs, symptoms, and triggers; (b) learning skills to manage symptoms, including PEF meter score interpretation, communication with adults (e.g. teachers, coaches, family members), medication use and MDI technique; (c) evaluating asthma symptoms and the effectiveness of management; and (d) discussing how to stay active in a safe manner] are covered as those in the asthma in-school classes.
  Asthma Day Camp
- Health Promotion In-school Class: The mock comparison follows the in-school format of 16 15-minute sessions; scheduled 3 sessions/week. The content is provided by trained health educators and includes skills practice (i.e., handwashing and brushing teeth) and health promotion topics of nutrition, healthy snacks, preventing colds, and safe exercise.
  Health Promotion in-school class
Period: Overall Study
Arm/Group | Asthma In-school Class | Asthma Day Camp | Health Promotion In-school Class
Started | 96 | 96 | 100
Completed | 84 | 89 | 81
Not Completed | 12 | 7 | 19
Not completed — Withdrawal by Subject | 12 | 7 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Asthma In-school Class | Asthma Day Camp | Health Promotion In-school Class | Total
Number analyzed (Participants) | 96 | 96 | 100 | 292
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 96 | 96 | 100 | 292
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.77 (1.25) | 8.83 (1.21) | 8.86 (1.29) | 8.82 (1.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 37 | 26 | 106
  Male | 53 | 59 | 74 | 186
Region of Enrollment [Number; unit: participants]
  United States | 96 | 96 | 100 | 292

OUTCOME MEASURES:

1. Primary Outcome: Absenteeism, End of Study
Description: (Days absent/days enrolled)x100 = absenteeism. Using data provided by the school district at the end of the study year.
Time Frame: 12 months
Population: Data for days enrolled and days absent was obtained from the school districts. Two school districts declined to provide the requested information, therefore there was substantial missing data for this variable.
Measure: Mean (Standard Deviation); unit: percentage of days enrolled
Arm/Group | Asthma In-school Class | Asthma Day Camp | Health Promotion In-school Class
Number analyzed (Participants) | 64 | 42 | 66
percentage of days enrolled | 3.83 (3.53) | 4.41 (4.04) | 3.68 (3.17)

2. Primary Outcome: Quality of Life, End of Study
Description: Self reported asthma-related quality of life. Outcome data were collected at end of study (Time 4). The Pediatric Asthma Quality of Life scale. Minimum score 23 to maximum score of 115. A higher score indicates worse quality of life. Mean scale scores are computed.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Asthma In-school Class | Asthma Day Camp | Health Promotion In-school Class
Number analyzed (Participants) | 84 | 89 | 82
units on a scale | 43.57 (15.40) | 43.87 (16.83) | 50.24 (20.76)

3. Primary Outcome: Number of Days Hospitalized, During Study Year
Description: Number of days hospitalized for asthma. Data were obtained from parent report at the second, third, and fourth data collection point. The number of hospitalization days were summed for a total number at the end of the 12 months.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: days hospitalized
Arm/Group | Asthma In-school Class | Asthma Day Camp | Health Promotion In-school Class
Number analyzed (Participants) | 81 | 89 | 84
days hospitalized | .04 (.19) | .09 (.51) | .26 (1.19)

4. Primary Outcome: Emergency Department Visits, Study Year
Description: Number of visits to Emergency Department for asthma. Data is obtained from parents at three time points (time 2, 3, and 4) and summed for total number of visits to the emergency department for asthma during the study year.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: number of visits
Arm/Group | Asthma In-school Class | Asthma Day Camp | Health Promotion In-school Class
Number analyzed (Participants) | 81 | 89 | 83
number of visits | .22 (.96) | .09 (.51) | .29 (.76)

5. Secondary Outcome: Asthma Self-management, Time 4
Description: Child self-report of asthma preventive and management activities, collected at each of 4 time points. This is the Time 4, final measure. Asthma Inventory for Children, 18-item scale, response scale 1-5, minimum score = 18, maximum score = 65, higher score = more frequent asthma self management behaviors.
Time Frame: Time 4, at 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Asthma In-school Class | Asthma Day Camp | Health Promotion In-school Class
Number analyzed (Participants) | 84 | 89 | 83
units on a scale | 51.84 (10.29) | 51.65 (9.09) | 51.44 (10.25)

6. Secondary Outcome: Home Asthma Management, Time 4, End of Study
Description: Parent report of asthma preventive and treatment activities. Data collected at final study visit, Time 4. Home Asthma Management scale, asthma preventive and asthma treatment behaviors performed by parent, response scale 1-5, scale range 16-70, higher scores = more frequent home asthma management behaviors.
Time Frame: Time 4 at 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Asthma In-school Class | Asthma Day Camp | Health Promotion In-school Class
Number analyzed (Participants) | 84 | 89 | 84
units on a scale | 61.16 (13.11) | 65.06 (13.51) | 62.34 (13.31)

7. Secondary Outcome: Metered Dose Inhaler Skill, Time 4
Description: Observation score of child's skill in using a placebo metered dose inhaler (a teaching inhaler). Observation data recorded by trained data collectors. 8-item scale listing the steps to perform proper inhalation technique. Number of correct steps are summed. Higher score = better skill in using inhaler. Collected at final, time 4 data visit.
Time Frame: Time 4 at 12 months
Measure: Mean (Standard Deviation); unit: number of correct steps
Arm/Group | Asthma In-school Class | Asthma Day Camp | Health Promotion In-school Class
Number analyzed (Participants) | 81 | 87 | 81
number of correct steps | 6.26 (1.37) | 6.30 (1.10) | 5.38 (1.34)

8. Secondary Outcome: Medication Adherence, Time 4
Description: Parent report of their child remembering/forgetting to take medications. 4-item scale (forgot to take medicine, was careless in taking medicine, stopped taking medicine due to feeling better, stopped taking medicine due to feeling worse), dichotomous response scale (yes, no), sum of number of yes items. Range 0-4, higher score means worse adherence. Data are collected at final data point, Time 4.
Time Frame: Time 4 at 12 months
Measure: Mean (Standard Deviation); unit: number of yes responses
Arm/Group | Asthma In-school Class | Asthma Day Camp | Health Promotion In-school Class
Number analyzed (Participants) | 84 | 88 | 84
number of yes responses | 0.74 (0.82) | 0.72 (0.84) | 0.81 (0.90)

9. Other Pre Specified Outcome: Lung Inflammation, Time 4
Description: Exhaled breath condensation collected and sent for lab analysis of NO3. Data collected at Time 4 visit. Higher values represent greater airway inflammation.
Time Frame: Time 4 at 12 months
Measure: Mean (Standard Deviation); unit: uM
Arm/Group | Asthma In-school Class | Asthma Day Camp | Health Promotion In-school Class
Number analyzed (Participants) | 82 | 83 | 82
uM | 1.93 (3.86) | 2.05 (4.53) | 1.97 (3.06)

10. Primary Outcome: Number of Asthma Hospitalizations Pre-Study Year
Description: Number of times hospitalized for asthma. Data is obtained from parents for the pre-study year for the previous 12 months.
Time Frame: 12 months before baseline
Measure: Mean (Standard Deviation); unit: number of hospitalizations
Arm/Group | Asthma In-school Class | Asthma Day Camp | Health Promotion In-school Class
Number analyzed (Participants) | 96 | 95 | 100
number of hospitalizations | 0.32 (1.53) | 0.15 (0.67) | 0.26 (0.84)

11. Primary Outcome: Absenteeism Pre-study Year
Description: (Days absent/days enrolled)x100 = absenteeism. Using data for the 12 months prior to study enrollment as the pre-study year. Data is provided by the participating school districts.
Time Frame: 12 months before baseline
Population: Data for days enrolled and days absent for the pre-study year was obtained from the school districts. Two school districts declined to provide the requested information, therefore there was substantial missing data for this variable.
Measure: Mean (Standard Deviation); unit: percentage of days enrolled
Arm/Group | Asthma In-school Class | Asthma Day Camp | Health Promotion In-school Class
Number analyzed (Participants) | 62 | 37 | 50
percentage of days enrolled | 3.17 (2.73) | 4.34 (3.20) | 4.00 (4.14)

12. Primary Outcome: Number of Days in Hospital for Asthma, Pre-Study Year
Description: Number of days hospitalized for asthma. Data is obtained from parents for the pre-study year for the previous 12 months.
Time Frame: 12 months before baseline
Measure: Mean (Standard Deviation); unit: days hospitalized
Arm/Group | Asthma In-school Class | Asthma Day Camp | Health Promotion In-school Class
Number analyzed (Participants) | 96 | 95 | 100
days hospitalized | 0.32 (1.53) | 0.15 (0.67) | 0.26 (0.84)

13. Primary Outcome: Number of Asthma Hospital Stays, During Study Year
Description: Number of hospital admissions for asthma. Data were obtained from parent report at the second, third, and fourth data collection point. The number of hospitalizations were summed for a total number at the end of the 12 months.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: number of hospital stays
Arm/Group | Asthma In-school Class | Asthma Day Camp | Health Promotion In-school Class
Number analyzed (Participants) | 80 | 89 | 84
number of hospital stays | 0.04 (0.19) | 0.06 (0.28) | 0.10 (0.30)

14. Primary Outcome: Emergency Department Visits, Pre-study Year
Description: Number of visits to Emergency Department for asthma. Data is obtained from parents for the pre-study year for the previous 12 months.
Time Frame: 12 months before baseline
Measure: Mean (Standard Deviation); unit: number of visits
Arm/Group | Asthma In-school Class | Asthma Day Camp | Health Promotion In-school Class
Number analyzed (Participants) | 96 | 96 | 100
number of visits | 0.42 (0.97) | 0.49 (1.13) | 0.76 (1.42)

15. Primary Outcome: Quality of Life, Pre-study Year
Description: Self reported asthma-related quality of life. Data were collected at study enrollment (time 1). The Pediatric Asthma Quality of Life scale. Minimum score 23 to maximum score of 115. A higher score indicates worse quality of life. Mean scale scores are computed.
Time Frame: 12 months before baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Asthma In-school Class | Asthma Day Camp | Health Promotion In-school Class
Number analyzed (Participants) | 96 | 96 | 100
units on a scale | 51.16 (18.98) | 53.57 (18.59) | 55.06 (21.65)

16. Secondary Outcome: Asthma Self-management, Time 3
Description: Child self-report of asthma preventive and management activities, collected at each of 4 time points. This is the Time 3 measure. Asthma Inventory for Children, 18-item scale, response scale 1-5, minimum score = 18, maximum score = 65, higher score = more frequent asthma self management behaviors.
Time Frame: Time 3 at 9 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Asthma In-school Class | Asthma Day Camp | Health Promotion In-school Class
Number analyzed (Participants) | 81 | 89 | 85
units on a scale | 51.60 (10.45) | 51.84 (9.27) | 52.58 (10.02)

17. Secondary Outcome: Asthma Self-management, Time 2
Description: Child self-report of asthma preventive and management activities, collected at each of 4 time points. This is the Time 2 measure. Asthma Inventory for Children, 18-item scale, response scale 1-5, minimum score = 18, maximum score = 65, higher score = more frequent asthma self management behaviors.
Time Frame: Time 2 at 5 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Asthma In-school Class | Asthma Day Camp | Health Promotion In-school Class
Number analyzed (Participants) | 86 | 91 | 89
units on a scale | 50.46 (10.44) | 51.01 (9.17) | 51.70 (9.11)

18. Secondary Outcome: Asthma Self-management, Time 1, Baseline
Description: Child self-report of asthma preventive and management activities, collected at each of 4 time points. This is the baseline, Time 1 measure. Asthma Inventory for Children, 18-item scale, response scale 1-5, minimum score = 18, maximum score = 65, higher score = more frequent asthma self management behaviors.
Time Frame: Time 1, baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Asthma In-school Class | Asthma Day Camp | Health Promotion In-school Class
Number analyzed (Participants) | 96 | 96 | 100
units on a scale | 48.57 (9.65) | 48.12 (8.95) | 50.45 (9.23)

19. Secondary Outcome: Home Asthma Management, Time 1, Baseline
Description: Parent report of asthma preventive and treatment activities. Data are collected at study enrollment, Time 1, baseline visit. Home Asthma Management scale, asthma preventive and asthma treatment behaviors performed by parent, response scale 1-5, scale range 16-70, higher scores = more frequent home asthma management behaviors.
Time Frame: Time 1, baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Asthma In-school Class | Asthma Day Camp | Health Promotion In-school Class
Number analyzed (Participants) | 96 | 96 | 100
units on a scale | 53.39 (10.96) | 53.07 (10.11) | 55.37 (9.18)

20. Secondary Outcome: Home Asthma Management, Time 2.
Description: Parent report of asthma preventive and treatment activities. Data collected at the time 2 visit. Home Asthma Management scale, asthma preventive and asthma treatment behaviors performed by parent, response scale 1-5, scale range 16-70, higher scores = more frequent home asthma management behaviors.
Time Frame: Time 2 at 5 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Asthma In-school Class | Asthma Day Camp | Health Promotion In-school Class
Number analyzed (Participants) | 86 | 91 | 89
units on a scale | 61.08 (21.37) | 61.60 (11.60) | 64.57 (18.06)

21. Secondary Outcome: Home Asthma Management, Time 3
Description: Parent report of asthma preventive and treatment activities. Data collected at third time point (Time 3). Home Asthma Management scale, asthma preventive and asthma treatment behaviors performed by parent, response scale 1-5, scale range 16-70, higher scores = more frequent home asthma management behaviors.
Time Frame: Time 3 at 9 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Asthma In-school Class | Asthma Day Camp | Health Promotion In-school Class
Number analyzed (Participants) | 81 | 89 | 85
units on a scale | 60.82 (12.56) | 64.41 (10.79) | 64.16 (11.50)

22. Secondary Outcome: Metered Dose Inhaler Skill, Time 3
Description: Observation score of child's skill in using a placebo metered dose inhaler (a teaching inhaler). Observation data recorded by trained data collectors. 8-item scale listing the steps to perform proper inhalation technique. Number of correct steps are summed. Higher score = better skill in using inhaler. Collected at time 3 data visit.
Time Frame: Time 3 at 9 months
Measure: Mean (Standard Deviation); unit: number of correct steps
Arm/Group | Asthma In-school Class | Asthma Day Camp | Health Promotion In-school Class
Number analyzed (Participants) | 80 | 85 | 84
number of correct steps | 6.16 (1.55) | 6.25 (1.24) | 5.63 (1.55)

23. Secondary Outcome: Metered Dose Inhaler Skill, Time 2
Description: Observation score of child's skill in using a placebo metered dose inhaler (a teaching inhaler). Observation data recorded by trained data collectors. 8-item scale listing the steps to perform proper inhalation technique. Number of correct steps are summed. Higher score = better skill in using inhaler. Collected at final, time 2 data visit.
Time Frame: Time 2 at 5 months
Measure: Mean (Standard Deviation); unit: number of correct steps
Arm/Group | Asthma In-school Class | Asthma Day Camp | Health Promotion In-school Class
Number analyzed (Participants) | 84 | 89 | 87
number of correct steps | 6.48 (1.18) | 6.20 (1.25) | 5.26 (1.39)

24. Secondary Outcome: Metered Dose Inhaler Skill, Time 1
Description: Observation score of child's skill in using a placebo metered dose inhaler (a teaching inhaler). Observation data recorded by trained data collectors. 8-item scale listing the steps to perform proper inhalation technique. Number of correct steps are summed. Higher score = better skill in using inhaler. Collected at enrollment visit, Time 1 data visit.
Time Frame: Time 1 at baseline
Measure: Mean (Standard Deviation); unit: number of correct steps
Arm/Group | Asthma In-school Class | Asthma Day Camp | Health Promotion In-school Class
Number analyzed (Participants) | 94 | 92 | 98
number of correct steps | 4.84 (1.60) | 4.87 (1.54) | 5.02 (1.46)

25. Secondary Outcome: Medication Adherence, Time 1
Description: Parent report of their child remembering/forgetting to take medications. 4-item scale (forgot to take medicine, was careless in taking medicine, stopped taking medicine due to feeling better, stopped taking medicine due to feeling worse), dichotomous response scale (yes, no), sum of number of yes items. Range 0-4, higher score means worse adherence. Data are collected at study enrollment, Time 1.
Time Frame: Time 1 at baseline
Measure: Mean (Standard Deviation); unit: number of yes responses
Arm/Group | Asthma In-school Class | Asthma Day Camp | Health Promotion In-school Class
Number analyzed (Participants) | 93 | 94 | 95
number of yes responses | 1.07 (1.04) | 1.07 (1.06) | 1.19 (1.13)

26. Secondary Outcome: Medication Adherence, Time 2
Description: Parent report of their child remembering/forgetting to take medications. 4-item scale (forgot to take medicine, was careless in taking medicine, stopped taking medicine due to feeling better, stopped taking medicine due to feeling worse), dichotomous response scale (yes, no), sum of number of yes items. Range 0-4, higher score means worse adherence. Data are collected at Time 2 visit.
Time Frame: Time 2 at 5 months
Measure: Mean (Standard Deviation); unit: number of yes responses
Arm/Group | Asthma In-school Class | Asthma Day Camp | Health Promotion In-school Class
Number analyzed (Participants) | 81 | 90 | 89
number of yes responses | 1.01 (1.07) | 0.87 (0.94) | 1.06 (1.10)

27. Secondary Outcome: Medication Adherence, Time 3
Description: Parent report of their child remembering/forgetting to take medications. 4-item scale (forgot to take medicine, was careless in taking medicine, stopped taking medicine due to feeling better, stopped taking medicine due to feeling worse), dichotomous response scale (yes, no), sum of number of yes items. Range 0-4, higher score means worse adherence. Data are collected at Time 3 visit.
Time Frame: Time 3 at 9 months
Measure: Mean (Standard Deviation); unit: number of yes responses
Arm/Group | Asthma In-school Class | Asthma Day Camp | Health Promotion In-school Class
Number analyzed (Participants) | 78 | 89 | 84
number of yes responses | 1.03 (1.02) | 0.89 (0.91) | 0.81 (0.98)

28. Other Pre Specified Outcome: Lung Inflammation, Time 1
Description: Exhaled breath condensation collected and sent for lab analysis of NO3. Data collected at Time 1 visit. Higher values represent greater airway inflammation.
Time Frame: Time 1 at baseline
Measure: Mean (Standard Deviation); unit: uM
Arm/Group | Asthma In-school Class | Asthma Day Camp | Health Promotion In-school Class
Number analyzed (Participants) | 92 | 93 | 99
uM | 1.69 (2.11) | 2.19 (2.50) | 2.03 (3.63)

29. Other Pre Specified Outcome: Lung Inflammation, Time 2
Description: Exhaled breath condensation collected and sent for lab analysis of NO3. Data collected at Time 2 visit. Higher values represent greater airway inflammation.
Time Frame: Time 2 at 5 months
Measure: Mean (Standard Deviation); unit: uM
Arm/Group | Asthma In-school Class | Asthma Day Camp | Health Promotion In-school Class
Number analyzed (Participants) | 84 | 85 | 88
uM | 1.91 (2.25) | 2.51 (3.20) | 2.11 (2.56)

30. Other Pre Specified Outcome: Lung Inflammation, Time 3
Description: Exhaled breath condensation collected and sent for lab analysis of NO3. Data collected at Time 3 visit. Higher values represent greater airway inflammation.
Time Frame: Time 3 at 9 months
Measure: Mean (Standard Deviation); unit: uM
Arm/Group | Asthma In-school Class | Asthma Day Camp | Health Promotion In-school Class
Number analyzed (Participants) | 80 | 86 | 83
uM | 1.83 (3.04) | 2.50 (3.32) | 2.61 (3.77)

ADVERSE EVENTS:
Time Frame: Every 3 months for up to 12 months
Arm/Group | Asthma In-school Class | Asthma Day Camp | Health Promotion In-school Class
Serious Adverse Events (participants affected / at risk) | 1/96 | 0/96 | 1/100
Other Adverse Events (participants affected / at risk) | 0/96 | 0/96 | 0/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Asthma In-school Class (N=96) | Asthma Day Camp (N=96) | Health Promotion In-school Class (N=100)
Hospital stay > 24 hours (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) — child was hospitalized for greater than 24 hours to manage asthma episode

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No